CLINICAL TRIAL: NCT07256847
Title: Effect of 6-Week High Intensity Interval Training on VO2max, Physical Competence and Sleep Quality in Sedentary Male University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ma Ruisi (Other)
Responsible Party: Sponsor-Investigator, Ma Ruisi, Co-Investigator, Jinan University Guangzhou
Organization: Jinan University Guangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBRE-23-0914
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2024-07

CONDITIONS: Sedentary Students; University Students
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (HIIT) group (Experimental): A 6-week HIIT exercise plan (running). Duration: Each session consists of 10 x 1-minute high-intensity bouts interspersed with 10 x 1-minute recovery periods. Adding the 3-minute warmup and 3-minute cool-down, each session totals approximately 26 minutes. This protocol is followed for 6 weeks.
  Intensity: High-intensity bouts are performed at 80-90% of HRmax (RPE 15-18). Recovery periods are at 40-50% of HRmax (RPE 11-13). Warm-up and cool-down are at 50% HRmax (RPE 11-13).
  Modality: Running, jogging, or brisk walking, either on a treadmill or outdoors.
  Supervision: The first three sessions are supervised in a laboratory setting. Subsequent sessions are unsupervised and performed at home with heart rate monitoring and remote data tracking via Polar Flow for Coach.
  Interventions: Other: High intensity interval training
- Control (No Intervention): Keep the usual life style without intervention.

INTERVENTIONS:
Other: High intensity interval training — A 6-week HIIT exercise plan (running). Duration: Each session consists of 10 x 1-minute high-intensity bouts interspersed with 10 x 1-minute recovery periods. Adding the 3-minute warmup and 3-minute cool-down, each session totals approximately 26 minutes. This protocol is followed for 6 weeks.
  Intensity: High-intensity bouts are performed at 80-90% of HRmax (RPE 15-18). Recovery periods are at 40-50% of HRmax (RPE 11-13). Warm-up and cool-down are at 50% HRmax (RPE 11-13).
  Modality: Running, jogging, or brisk walking, either on a treadmill or outdoors. Supervision: The first three sessions are supervised in a laboratory setting. Subsequent sessions are unsupervised and performed at home with heart rate monitoring and remote data tracking via Polar Flow for Coach.
  Arms: High-intensity interval training (HIIT) group

SUMMARY:
This study aims to investigate the effects of a 6-week high-intensity interval training (HIIT) intervention on physical fitness, cardiorespiratory capacity (VO2max), and sleep quality among sedentary male college students. Through a randomized controlled trial, we seek to examine whether HIIT, as a time-efficient exercise modality, can effectively improve these health-related outcomes in young adults who maintain predominantly sedentary lifestyles. This research will provide evidence-based insights into the effectiveness of HIIT as a potential intervention strategy to address the physical and physiological consequences of prolonged sitting behavior among university students.

ELIGIBILITY:
Inclusion Criteria:

1. university students;
2. daily sedentary time > 8 hours;
3. healthy individuals who are capable of physical tests or HIIT;
4. no regular exercise habits;
5. can understand English or Chinese.

Exclusion Criteria:

1. self-reported history of neurological, psychiatric, or medical diseases;
2. current intake of medications and/or recreational drugs that could affect the central nervous system and/or the ability to learn.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — To control for sex-specific variations in exercise responses, this study was only restricted to biological male university students.
Enrollment: 56 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
VO2max | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Progressive Aerobic Cardiovascular Endurance Run 20-m (measured in laps)
Sleep Quality | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Pittsburgh Sleep Quality Index (PSQI) (scored from 0 to 21, with higher scores indicating worse sleep quality)
Handgrip | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Handgrip dynamometer (measured in kilograms)
Core strength | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Plank test (measured in second)
Balance | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Unipedal stance test (measured in second)
Agility | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Agility T-test (measured in second)
Flexibility | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Sit and Reach Test
Body composition (measured in centimeter) | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Bioelectrical impedance analysis (BIA) device (MC-780MA)

OTHER OUTCOMES:
Carbohydrate Intake | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Daily carbohydrate consumption measured by validated 3-day food diary (measured in grams/day)
Fat Intake | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Daily fat consumption measured by a validated 3-day food diary (measured in grams/day)
Protein Intake | Baseline (pre-intervention) and immediately after 6-week intervention completion
  Daily protein consumption measured by a validated 3-day food diary (measured in grams/day)
Physical Activity Level | Baseline (pre-intervention) and immediately after 6-week intervention completion
  International Physical Activity Questionnaire (IPAQ) long form (measured in MET-minutes/week, range: 0 to no upper limit, with higher scores indicating higher levels of physical activity)

CONTACTS AND LOCATIONS:
Locations (1):
- SSPE, The Chinese University of Hong Kong, Hong Kong, None Selected, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yano A, Hidaka E, Fujiwara K, Iimoto M. Induction of primary root curvature in radish seedlings in a static magnetic field. Bioelectromagnetics. 2001 Apr;22(3):194-9. doi: 10.1002/bem.38. PMID 11255215
- [Background] Eather N, Riley N, Miller A, Smith V, Poole A, Vincze L, Morgan PJ, Lubans DR. Efficacy and feasibility of HIIT training for university students: The Uni-HIIT RCT. J Sci Med Sport. 2019 May;22(5):596-601. doi: 10.1016/j.jsams.2018.11.016. Epub 2018 Nov 24. PMID 30509862